CLINICAL TRIAL: NCT05714501
Title: Millipede AspiRation for Revascularization in Stroke (MARRS) Study
Acronym: MARRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perfuze (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN040
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single Arm (Experimental): Millipede System
  Interventions: Device: Millipede System

INTERVENTIONS:
Device: Millipede System — Mechanical thrombectomy

SUMMARY:
The objectives of the study are to examine the performance and safety characteristics of the Millipede System when used for revascularization of patients with acute ischemic stroke due to Large Vessel Occlusions (LVOs) and to record associated clinical outcomes.

DETAILED DESCRIPTION:
Ischemic stroke is a life-threatening condition. Annually, approximately 795,000 people in the United States have a stroke.

The MARRS study is an interventional, open label, single arm, multi center, prospective clinical investigation. The objectives of the study are to evaluate the performance and safety characteristics of the Millipede System in patients presenting with acute ischemic stroke due to LVOs and to record clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥ 18 and ≤ 85 years.
2. Pre-stroke mRS score of ≤ 1.
3. Baseline NIHSS score of ≥ 6.
4. A new focal disabling neurologic deficit consistent with acute cerebral ischemia.
5. Evidence of a large vessel occlusion of the intracranial ICA (including T or L occlusions), the M1 or M2 segments of the MCA, the intracranial vertebral artery, or the basilar artery on magnetic resonance angiography (MRA) or computed tomography angiography (CTA).
6. Subject belongs to one of the following subgroups:

   1. Subject is ineligible for thrombolytic therapy, OR
   2. Subject is eligible for thrombolytic therapy and thrombolytic therapy was administered without delay and per current practice guidelines.
7. For strokes in the anterior circulation, the following imaging criteria should be met:

   1. Magnetic Resonance Imaging (MRI) criterion: volume of diffusion restriction visually assessed as ≤ 50 mL, or Alberta Stroke Program Early CT Score (ASPECTS) 6-10; OR
   2. Computed Tomography (CT) criterion: Alberta Stroke Program Early CT Score (ASPECTS) 6-10 on baseline CT or Computed Tomography Angiography (CTA)- source images, or volume of significantly lowered relative Cerebral Blood Flow (rCBF) <30% (volume of ≤ 50 mL if CT perfusion is performed).
8. For strokes in the posterior circulation, the following imaging criterion should be met: pcASPECTS score 8 to 10 on baseline CT, CTA-source images, or Diffusion- Weighted Imaging (DWI) MRI.
9. The interventionalist estimates that arterial puncture can be completed within 8 hours of onset/last known well.
10. Informed consent obtained in accordance with the applicable country-specific regulations and as approved by the IRB/ REC.
11. Angiographic confirmation of a single large vessel occlusion (mTICI of 0-1) of the intracranial ICA (including T or L occlusions), the M1 or M2 segments of the MCA, the intracranial vertebral artery, or the basilar artery that is accessible to the Millipede System.

Exclusion Criteria:

1. Known previous stroke within the past 3 months.
2. Females who are known to be pregnant or breastfeeding.
3. In the Investigator's opinion, any known comorbidity (including COVID-19) that may complicate treatment or prevent improvement or follow-up.
4. Subject currently participating in or has previously participated in another trial involving an investigational device or drug within 30 days of enrollment.
5. Known history of severe contrast allergy.
6. Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluation.
7. Life expectancy of less than 6 months prior to stroke onset.
8. Known cocaine use at time of treatment.
9. Known history of coagulation factor deficiency or oral anti-coagulant therapy with an International Normalized Ratio (INR) of more than 3.0.
10. Known history of treatment with heparin within 48 hours with a Partial Thromboplastin Time (PTT) more than two times the laboratory normal.
11. Known history of treatment with a direct thrombin inhibitor within 48 hours with a PTT more than 1.5 times the laboratory normal.
12. Known glucose level< 50 mg/dl (2.78 mmol/L) or > 400 mg/dl (22.20 mmol/L).
13. Known platelet count <50,000/µL.
14. Clinical history, past imaging or clinical judgement suggest that the intracranial occlusion is chronic.
15. For all patients, severe sustained hypertension with SBP >220 mmHg and/or DBP >120 mmHg; for patients treated with thrombolytic therapy, sustained hypertension despite treatment with SBP >185 mmHg and/or DBP > 110 mmHg.
16. Renal failure with serum creatinine ≥3 mg/dL or Glomerular Filtration Rate (GFR) <30 mL/min.
17. Ongoing seizure due to stroke.
18. Initially treated with intra-arterial thrombolytics or a different neurothrombectomy device before use of the Millipede System.
19. Clinical symptoms of bilateral stroke or stroke in multiple territories.
20. Known history of cerebral vasculitis.
21. Evidence of active systemic infection (e.g. septicemia). Exceptions: common cold, hepatitis B virus (HBV), hepatitis C virus (HCV).
22. Any known hemorrhagic or coagulation deficiency.
23. Evidence of current intracranial hemorrhage on imaging.
24. Significant mass effect with midline shift.
25. Known arterial condition in a proximal vessel that requires treatment or prevents access to the site of occlusion or safe recovery of the investigational device (for example, severe stenosis, complete occlusion in the cervical ICA, tandem occlusion).
26. Suspicion or evidence of aortic dissection, septic embolus, or bacterial endocarditis.
27. Evidence of dissection in the extracranial or intracranial cerebral arteries.
28. Excessive arterial tortuosity that may preclude device placement as determined by CTA/Magnetic Resonance Angiography (MRA) and/or conventional angiography.
29. Evidence of multiple vascular occlusions (e.g., bilateral anterior circulation, anterior/posterior circulation, concurrent occlusions in the anterior cerebral artery (ACA) and MCA, other concurrent ipsilateral occlusions in the same or different territories).
30. CT or MRI showing mass effect or intracranial tumor (apart from small meningioma, ≤ 2 cm in diameter).
31. Known cancer with metastases.
32. Known aneurysm at or near the target treatment segment.
33. Angiographic evidence of known or suspected underlying intracranial vasculopathy or atherosclerotic lesions responsible for the target occlusion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with successful reperfusion, defined as achieving a modified Thrombolysis in Cerebrovascular Infarction (mTICI) score of 2b or greater, after ≤3 passes with the Millipede System without additional therapy. | During procedure.
  mTICI of 2b or greater indicating successful reperfusion.
The safety of the Millipede System will be determined through a review of all adverse events (AEs) recorded during the study.post-procedure. | From Day 0 (procedure) through to the 90 Day visit.
  All AEs will be analyzed, with specific attention to the rate of all intracranial hemorrhage (ICH), including symptomatic intracranial hemorrhage (sICH), subarachnoid hemorrhage (SAH), non-hemorrhagic AEs capable of producing neurological deterioration, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Raul Nogueira, MD, Principal Investigator — University of Pittsburgh Medical Center (UPMC), Pittsburgh, USA; Marc Ribo, MD, Principal Investigator — Vall D'Hebron Hospital, Barcelona, Spain; Ricardo Hanel, MD, Principal Investigator — Baptist Health Research Institute, Jacksonville, USA
Locations (23):
- United States (15):
  - Yale University Hospital, New Haven, Connecticut
  - Baptist Health Research Institute, Jacksonville, Florida
  - Tampa General Hosital, Tampa, Florida
  - Emory, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University Of Rochester Medical Center (URMC), Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Mercy Health, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Semmes Murphey Foundation, Memphis, Tennessee
  - Valley Baptist Medical Center, Harlingen, Texas
  - UT Houston, Houston, Texas
- France (6):
  - CHU Bordeaux, Bordeaux, Bordeaux
  - CHU de Nantes - HGRL, Nantes, Nantes
  - CHRU Strasbourg, Strasbourg, Strasbourg
  - CHU Montpellier, Montpellier
  - CHRU de Nancy, Nancy
  - Toulouse University Hospital -CHU Purpan, Toulouse
- Spain (2):
  - Hospital Universitario La Paz, Madrid, Madrid
  - Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No